CLINICAL TRIAL: NCT00124735
Title: An Open-label, Randomized, Phase IIIB, Multicenter Trial to Evaluate the Pharmacodynamic Parameters of Intubation Bolus, and Bolus and Infusion Maintenance Doses of Zemuron® in Pediatric and Adolescent Subjects
Brief Title: A Study to Determine the Dose Requirements of Rocuronium Bromide (Zemuron®) in Pediatric and Adolescent Subjects (21048)(COMPLETED)(P05797)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05797; 21048
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2009-04-15 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rocuronium bolus maintenance (Experimental): Rocuronium bolus maintenance
  Interventions: Drug: Rocuronium bolus maintenance
- Rocuronium continuous infusion maintenance (Experimental): Rocuronium continuous infusion maintenance
  Interventions: Drug: rocuronium continuous infusion maintenance

INTERVENTIONS:
Drug: Rocuronium bolus maintenance — Subjects received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation
  Other Names: Zemuron; ORG 9426
  Arms: Rocuronium bolus maintenance
Drug: rocuronium continuous infusion maintenance — Subjects received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation
  Other Names: Zemuron; ORG 9426
  Arms: Rocuronium continuous infusion maintenance

SUMMARY:
The primary purpose of this study is to determine the dose requirements of rocuronium bromide when administered as a bolus dose (a single, large dose) for intubation (insertion of a tube through the nose or mouth into the trachea to provide artificial ventilation) and when administered by either continuous infusion or bolus doses for maintenance of muscle relaxation in term neonates (birth to <28 days old), infants (28 days to <=3 months) and toddlers (>3 months to <=2 years), children (2 years to less than or equal to 11 years of age), and adolescents (>11 years to less than or equal to 17 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects from birth up to 17 years of age who are scheduled for surgery with an anticipated duration of anesthesia of about 2 hours or more requiring a maintenance muscle relaxation dose(s).

Exclusion Criteria:

* Subjects whose parent(s) or legal guardian(s) are not willing to give written consent and where applicable, subjects who have not given appropriate assent to participate in the trials will not be allowed to enter.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2004-10; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

REFERENCES:
- [Result] Bhattacharya ST, Jeffrey Koh J, Martin L, Suresh S, Frietsch T. Randomized, Multicenter Trial of Rocuronium in Neonates, Infants, Toddlers, Children & Adolescents [abstract]. Anesthesiology. 2009;111(5):A841.

RESULTS

PARTICIPANT FLOW:
Groups:
- Rocuronium Bolus Maintenance - Neonate (BN): Neonate subjects that received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation
- Rocuronium Bolus Maintenance - Infants (BI): Infant subjects that received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation
- Rocuronium Bolus Maintenance - Toddlers (BT): Toddler subjects that received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation
- Rocuronium Bolus Maintenance -Children (BC): Children subjects that received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation
- Rocuronium Bolus Maintenance - Adolescents (BA): Adolescent subjects that received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation
- Rocuronium Continuous Infusion Maintenance - Neonates (IN): Neonate subjects that received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation
- Rocuronium Continuous Infusion Maintenance - Infants (II): Infant subjects that received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation
- Rocuronium Continuous Infusion Maintenance - Toddlers (IT): Toddler subjects that received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation
- Rocuronium Continuous Infusion Maintenance - Children (IC): Children subjects that received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation
- Rocuronium Continuous Infusion Maintenance - Adolescents (IA): Adolescent subjects that received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation
Period: Overall Study
Arm/Group | Rocuronium Bolus Maintenance - Neonate (BN) | Rocuronium Bolus Maintenance - Infants (BI) | Rocuronium Bolus Maintenance - Toddlers (BT) | Rocuronium Bolus Maintenance -Children (BC) | Rocuronium Bolus Maintenance - Adolescents (BA) | Rocuronium Continuous Infusion Maintenance - Neonates (IN) | Rocuronium Continuous Infusion Maintenance - Infants (II) | Rocuronium Continuous Infusion Maintenance - Toddlers (IT) | Rocuronium Continuous Infusion Maintenance - Children (IC) | Rocuronium Continuous Infusion Maintenance - Adolescents (IA)
Started | 5 | 8 | 18 | 21 | 19 | 7 | 6 | 20 | 25 | 20
Completed | 4 | 6 | 18 | 18 | 17 | 5 | 6 | 19 | 22 | 18
Not Completed | 1 | 2 | 0 | 3 | 2 | 2 | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocuronium Bolus Maintenance - Neonate (BN) | Rocuronium Bolus Maintenance - Infants (BI) | Rocuronium Bolus Maintenance - Toddlers (BT) | Rocuronium Bolus Maintenance -Children (BC) | Rocuronium Bolus Maintenance - Adolescents (BA) | Rocuronium Continuous Infusion Maintenance - Neonates (IN) | Rocuronium Continuous Infusion Maintenance - Infants (II) | Rocuronium Continuous Infusion Maintenance - Toddlers (IT) | Rocuronium Continuous Infusion Maintenance - Children (IC) | Rocuronium Continuous Infusion Maintenance - Adolescents (IA) | Total
Number analyzed (Participants) | 5 | 6 | 18 | 18 | 17 | 5 | 6 | 19 | 23 | 20 | 137
Age, Categorical [Count of Participants; unit: Participants] — Total of 137 subjects include all subjects who received rocuronium
  Participants
    <=18 years | 5 | 6 | 18 | 18 | 17 | 5 | 6 | 19 | 23 | 20 | 137
    Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Total of 137 subjects include all subjects who received rocuronium
  Participants
    Female | 2 | 1 | 1 | 8 | 6 | 2 | 3 | 6 | 11 | 12 | 52
    Male | 3 | 5 | 17 | 10 | 11 | 3 | 3 | 13 | 12 | 8 | 85

OUTCOME MEASURES:

1. Primary Outcome: Total Dose of Zemuron (Rocuronium) Administered
Description: Total dose from administration of intubating dose to reappearance of T3 (the third twitch of a Train of Four [TOF] stimulation) after the last maintenance bolus dose or discontinuation of Zemuron (rocuronium) infusion (Per protocol [PP] data set)
Time Frame: during surgery
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Rocuronium Bolus Maintenance - Neonate (BN) | Rocuronium Bolus Maintenance - Infants (BI) | Rocuronium Bolus Maintenance - Toddlers (BT) | Rocuronium Bolus Maintenance -Children (BC) | Rocuronium Bolus Maintenance - Adolescents (BA) | Rocuronium Continuous Infusion Maintenance - Neonates (IN) | Rocuronium Continuous Infusion Maintenance - Infants (II) | Rocuronium Continuous Infusion Maintenance - Toddlers (IT) | Rocuronium Continuous Infusion Maintenance - Children (IC) | Rocuronium Continuous Infusion Maintenance - Adolescents (IA)
Number analyzed (Participants) | 3 | 5 | 13 | 14 | 15 | 5 | 2 | 12 | 19 | 15
mg/kg | 0.91 (0.17) | 0.78 (0.07) | 0.86 (0.18) | 0.81 (0.10) | 0.96 (0.16) | 1.01 (0.37) | 0.84 (0.15) | 1.00 (0.25) | 1.26 (0.78) | 0.99 (0.37)

2. Secondary Outcome: Duration of Recovery of T4/T1 Ratio (TOF Fourth Twitch to First Twitch) 70%
Description: The time it takes for the the T4 to T1 ratio to reach 70%. The T4/T1 ratio is indicative of recovery. At complete recovery, the T4/T1 ratio is 1.0 (100%).
Time Frame: after surgery, from the reappearance of T3 after Zemuron(R) (rocuronium) infusion/last bolus dose of Zemuron(R) (rocuronium)
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rocuronium Bolus Maintenance - Neonate (BN) | Rocuronium Bolus Maintenance - Infants (BI) | Rocuronium Bolus Maintenance - Toddlers (BT) | Rocuronium Bolus Maintenance -Children (BC) | Rocuronium Bolus Maintenance - Adolescents (BA) | Rocuronium Continuous Infusion Maintenance - Neonates (IN) | Rocuronium Continuous Infusion Maintenance - Infants (II) | Rocuronium Continuous Infusion Maintenance - Toddlers (IT) | Rocuronium Continuous Infusion Maintenance - Children (IC) | Rocuronium Continuous Infusion Maintenance - Adolescents (IA)
Number analyzed (Participants) | 2 | 4 | 10 | 13 | 11 | 3 | 1 | 9 | 15 | 13
minutes | 29.62 (13.60) | 33.25 (16.17) | 22.65 (7.62) | 16.19 (6.70) | 28.04 (13.33) | 43.32 (1.53) | 33.25 (0.00) | 23.08 (13.40) | 18.37 (12.69) | 27.59 (12.51)

3. Secondary Outcome: Duration of Recovery of T4/T1 (TOF Fourth Twitch to First Twitch) Ratio 80%
Description: The time it takes for the the T4 to T1 ratio to reach 80%. The T4/T1 ratio is indicative of recovery. At complete recovery, the T4/T1 ratio is 1.0 (100%).
Time Frame: as for outcome 2
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rocuronium Bolus Maintenance - Neonate (BN) | Rocuronium Bolus Maintenance - Infants (BI) | Rocuronium Bolus Maintenance - Toddlers (BT) | Rocuronium Bolus Maintenance -Children (BC) | Rocuronium Bolus Maintenance - Adolescents (BA) | Rocuronium Continuous Infusion Maintenance - Neonates (IN) | Rocuronium Continuous Infusion Maintenance - Infants (II) | Rocuronium Continuous Infusion Maintenance - Toddlers (IT) | Rocuronium Continuous Infusion Maintenance - Children (IC) | Rocuronium Continuous Infusion Maintenance - Adolescents (IA)
Number analyzed (Participants) | 2 | 3 | 9 | 11 | 11 | 3 | 1 | 9 | 15 | 11
minutes | 36.62 (17.14) | 43.58 (21.47) | 32.39 (12.84) | 20.43 (9.79) | 35.75 (19.43) | 57.83 (12.33) | 44.75 (0.00) | 29.47 (16.65) | 21.82 (14.57) | 35.45 (17.02)

4. Secondary Outcome: Duration of Recovery of T4/T1 (TOF Fourth Twitch to First Twitch) Ratio 90%
Description: The time it takes for the the T4 to T1 ratio to reach 90%. The T4/T1 ratio is indicative of recovery. At complete recovery, the T4/T1 ratio is 1.0 (100%).
Time Frame: as for outcome 2
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rocuronium Bolus Maintenance - Neonate (BN) | Rocuronium Bolus Maintenance - Infants (BI) | Rocuronium Bolus Maintenance - Toddlers (BT) | Rocuronium Bolus Maintenance -Children (BC) | Rocuronium Bolus Maintenance - Adolescents (BA) | Rocuronium Continuous Infusion Maintenance - Neonates (IN) | Rocuronium Continuous Infusion Maintenance - Infants (II) | Rocuronium Continuous Infusion Maintenance - Toddlers (IT) | Rocuronium Continuous Infusion Maintenance - Children (IC) | Rocuronium Continuous Infusion Maintenance - Adolescents (IA)
Number analyzed (Participants) | 1 | 3 | 8 | 8 | 7 | 1 | 1 | 9 | 13 | 10
minutes | 28.25 (0) | 53.66 (14.58) | 45.31 (18.20) | 23.09 (10.90) | 49.25 (31.73) | 52.25 (0) | 50.75 (0) | 37.86 (18.46) | 28.02 (21.46) | 38.68 (16.08)

ADVERSE EVENTS:
Description: All subjects who received rocuronium were included in the safety analyses.
  Information regarding adverse events were obtained by questioning or examining the subject. At each visit during the treatment period, all new complaints and symptoms were recorded.
Groups:
- Rocuronium Bolus Maintenance: Subjects that received a bolus dose of rocuronium for intubation followed by bolus doses for maintenance of muscle relaxation (includes neonates, infants, toddlers, children, and adolescents).
- Rocuronium Continuous Infusion Maintenance: Subjects that received a bolus dose of rocuronium for intubation followed by continuous infusion of rocuronium for maintenance of muscle relaxation (includes neonates, infants, toddlers, children, and adolescents)
Arm/Group | Rocuronium Bolus Maintenance | Rocuronium Continuous Infusion Maintenance
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/73
Other Adverse Events (participants affected / at risk) | 10/64 | 9/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium Bolus Maintenance (N=64) | Rocuronium Continuous Infusion Maintenance (N=73)
postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium Bolus Maintenance (N=64) | Rocuronium Continuous Infusion Maintenance (N=73)
procedural pain (Injury, poisoning and procedural complications) | 10 (12) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to Organon, at least 6 weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.